CLINICAL TRIAL: NCT02238418
Title: Vitamin D Supplementation in Children and Adolescents Seen in the Paediatric Nephrology Service: Study of the Efficacy of Service Usual Care (Cholecalciferol) and Its Impact on Calciuria.
Brief Title: Efficacy of Usual Vitamin D Supplementation and Its Impact on Children and Adolescents Calciuria.
Acronym: VITATOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-812; 2013-002710-13 (EudraCT Number)
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease; Renal Transplantation; Nephrotic Syndrome
Keywords: Vitamin D, Calciuria, Paediatrics, Nephrology
MeSH Terms: conditions — Renal Insufficiency, Chronic; Nephrotic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Usual vitamin D supplementation (Experimental)
  Interventions: Drug: Cholecalciferol vial (100 000 UI)

INTERVENTIONS:
Drug: Cholecalciferol vial (100 000 UI) — VISIT 1:
  Patient > 60 kg and initial 25OHD serum concentration < 25nmol/L : prescription of 4 vials to be taken every 2 weeks between 25 and 50 nmol/L: prescription of 3 vials to be taken every 2 weeks between 50 and 75 nmol/L: prescription of 2 vials to be taken every 2 weeks Patient between 20 and 60 kg and initial 25OHD serum concentration < 25nmol/L: prescription of 2 vials to be taken every month between 25 and 50 nmol/L: prescription of 2 vials to be taken every 6 weeks between 50 and 75 nmol/L: prescription of 1 single vial Patient < 20 kg and initial 25OHD serum concentration < 75 nmol/L: prescription of 1 single vial
  A local lab will performed urinary dosage of calciuria and creatininuria:
  * at days 0, 1, 2, 3, 4 and 7 after the first intake of a 25OHD vial
  * at days 0, 2 and 4 after other intakes (when applicable)
  VISIT 2:
  25OHD serum concentration will then be dosed at month 2 after visit 1

SUMMARY:
Vitamin D is not seen anymore only as a phosphocalcic and bone hormone, but also as having an effect on global health (anti-infective, anti-inflammatory, anti-tumour roles and cardiovascular protection).

Until recently, vitamin D repletion was defined as the minimal concentration that enables the prevention of rickets in children and osteomalacia in adults, i.e, approximately 8 ng/mL (20 nmol/L). However, most of the international experts agree to set minimal threshold of 25 OH vitamin D serum concentration, higher than the one previously admitted, with a limit of 20 ng/mL (50 nmol/L) to define a vitamin D deficiency and a limit of 30 ng/mL (75 nmol/L) to define vitamin D insufficiency.

Recommendations for Vit D supplementation in healthy children were updated in France in 2012. The invariable supplementation of infants and toddlers is efficient since deficiency-related rickets have almost disappeared; however there is very few information in ill children populations.

Vit D supplementation tolerance is usually considered as good and over-dosage risks are low, however these studies were conducted more than 30 years ago, and as far as we know, there is no study about calcium urinary excretion kinetics after intake of a 100 000 IU vial of cholecalciferol (Uvedose®). When 25 OH vitamin D serum concentrations exceeds 200 ng/mL, which is very rare in daily practice, toxic effects of Vit D may theoretically be observed, particularly hypercalcemia and hypercalciuria.

Vitamin D deficit is very common in children with chronic kidney disease (CKD) with a 50 to 92% prevalence depending on the studies; it it is a risk factor for secondary hyperparathyroidism.

Although international guidelines regarding the care of CKD children recommend 25 OH vitamin D serum concentrations over 75 nmol/L, there are no practical recommendations in terms of dose and frequency of native Vit D treatment.

Therefore, the objectives of the present study has are the following:

* to validate prospectively the efficacy of our service usual care for Vit D supplementation of children and adolescents seen in the paediatric nephrology department.
* and to study the effect of Vit D supplementation (100 000 IU vial of cholecalciferol) on calciuria in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age : between [18 mo et 18 yo[
* Patients seen in the paediatric nephrology service and having :

  * Chronic kidney disease
  * Renal transplant
  * Stable nephrotic syndrome (i.e., normal protidemia at inclusion)
* Initial 25 OH vitamin D concentration < 75nmol/l
* Patient agree to participate (if old enough to give his agreement) and written informed consent signed by parents
* Patients affiliated within the French universal healthcare system

Exclusion Criteria:

- Contraindication to 100 000 IU Uvedose® treatment (according to the Summary of Product Characteristics: known hypersensitivity to vitamin D or hypercalcemia, hypercalciuria or nephrolithiasis).

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of usual vitamin D supplementation | Day 60
  The 25 OH vitamin D serum concentration will be measured at inclusion (before treatment intake) and 2 months after supplementation. No extra blood intake is programmed since this parameter is always measured in this population. The main evaluation criterion is defined as a 25 OH vitamin D serum concentration over 75 nmol/l at month 2. This defines the success of supplementation. The failure is defined as a 25 OH vitamin D serum concentration under 75 nmol/l at month 2.

SECONDARY OUTCOMES:
Kinetics of calciuria after a 100 000 IU vial of cholecalciferol | Day 0, day 1, day 2, day 3, day 4, day 7 after treatment intake.
  Calciuria (absolute and normalized with the calculation of the ratio urinary calcium/creatinine) will be measured on the first morning urine at those time points after each vial intake. Measurements will be made in the unique local laboratory chosen by each patient. Thus the lab will be different between patients but must remain the same for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Justine Bacchetta, MD, Principal Investigator — HCL
Locations (1):
- Centre de Référence des Maladies Rénales Rares - Hospices Civils de Lyon - Service de Néphrologie et Rhumatologie Pédiatriques - Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aurelle M, Basmaison O, Ranchin B, Kassai-Koupai B, Sellier-Leclerc AL, Bertholet-Thomas A, Bacchetta J. Intermittent cholecalciferol supplementation in children and teenagers followed in pediatric nephrology: data from a prospective single-center single-arm open trial. Eur J Pediatr. 2020 Apr;179(4):661-669. doi: 10.1007/s00431-019-03553-y. Epub 2019 Dec 24. PMID 31873802